CLINICAL TRIAL: NCT07264634
Title: A Study to Assess the Amount of Palopegteriparatide in Breast Milk of Lactating Females Requiring YORVIPATH® (Palopegteriparatide)
Status: Not yet recruiting | Type: Observational
Sponsor: Ascendis Pharma A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: ASND0044
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Palopegteriparatide: Pregnant women exposed to palopegteriparatide during pregnancy
  Interventions: Drug: Palopegteriparatide

INTERVENTIONS:
Drug: Palopegteriparatide — Palopegteriparatide prescribed as per normal clinical practice

SUMMARY:
This is an observational, opportunistic lactation study to be conducted in lactating female participants who are currently receiving therapeutic doses of YORVIPATH as part of their usual care and who have chosen to breastfeed their infant(s). The potential transfer of palopegteriparatide into breast milk will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Lactating female participants 18 years of age or older treated with YORVIPATH as part of their usual medical care and who have chosen to breastfeed. Note: The participant must have been taking YORVIPATH for a minimum of 14 days prior to sample collection.
* 2. The major source of infant nutrition must be breast milk (Note: Only one supplemental bottle of no more than up to 8 oz of formula per day will be allowed during the 14 days before start of the study).
* 3. Daily dose of YORVIPATH administered within the last 14 days has been stable.
* 4. Participants recruited from other sources must enroll in the Pregnancy Registry before being allowed to participate in the Lactation Study.
* 5. Written consent or eConsent obtained.

Exclusion Criteria:

* 1. Presence of any medical condition that, in the opinion of the investigator, may impair the ability to breastfeed during this study, including but not limited to mastitis and nipple malformation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Eligible females will be actively recruited from the US participants in the pregnancy registry. Females in the US who want to participate in the lactation study must first enroll in the pregnancy registry and meet the lactation study eligibility criteria study to participate. Females may self enroll into the study or may be enrolled by their healthcare provider (HCP).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the transfer of palopegteriparatide into human breast milk of lactating female participants who are breastfeeding while being treated with YORVIPATH | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Ascendis Pharma A/S